CLINICAL TRIAL: NCT05009511
Title: MRI Markers of Feedback Timing During Learning in Individuals with TBI with and Without Clinical Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Moss Rehabilitation Research Institute (Other)
Responsible Party: Principal Investigator, Ekaterina Dobryakova, Principal Investigator, Kessler Foundation
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: R-1142-21; R01NS121107 (NIH)
Record Dates: First submitted 2021-07-30; First posted 2021-08-17 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2023-12

CONDITIONS: Traumatic Brain Injury; Major Depressive Disorder
Keywords: fMRI; Traumatic Brain Injury; Major Depressive Disorder; Learning; Memory; Feedback; Rehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Traumatic Brain Injury (TBI) (Experimental): Individuals with moderate-to-severe injury severity, defined as post-traumatic amnesia lasting more than 24hrs, loss of consciousness lasting more than 30 min, Glasgow Coma Scale (GCS) score less than 13.
  Interventions: Behavioral: Learning through feedback
- Traumatic Brain Injury (TBI) with MDD (Experimental): Individuals with moderate-to-severe injury severity, defined as post-traumatic amnesia lasting more than 24hrs, loss of consciousness lasting more than 30 min, Glasgow Coma Scale (GCS) score less than 13. In addition, individuals will have a diagnosis of major depressive disorder (MDD) as per DSM-5.
  Interventions: Behavioral: Learning through feedback
- Major Depressive Disorder (MDD) (Experimental): Individuals meeting criteria for major depressive disorder (MDD) including qualifiers 'in partial remission' or 'in full remission' if they are actively in treatment for the condition and still carry the depression diagnosis.
  Interventions: Behavioral: Learning through feedback
- Healthy Individuals (Experimental): Healthy individuals without psychiatric and neurological conditions.
  Interventions: Behavioral: Learning through feedback

INTERVENTIONS:
Behavioral: Learning through feedback — The goal of this investigation is to examine the influence of feedback timing on learning and brain function.

SUMMARY:
The goal of this proposal is to examine the influence of feedback timing on learning and brain function in individuals with moderate-to-severe traumatic brain injury (TBI), with and without depression.

DETAILED DESCRIPTION:
The overall objective of the proposed project is to investigate brain mechanisms during learning in individuals with traumatic brain injury (TBI) with and without clinical depression. Such knowledge can help guide rehabilitation strategies and reduce the burden of TBI. Feedback about the accuracy of one's actions can improve learning by informing an individual whether his/her action is correct or not. Individuals with depression have been shown to have learning deficits and altered brain activity during learning compared to healthy individuals when feedback is presented immediately. Impaired learning through immediate feedback has also been observed in Parkinson's disease (PD) patients. However, PD patients are able to learn from feedback when it is presented after a delay, engaging separate neural mechanisms. Individuals with TBI have also been shown to have learning deficits that are likely exacerbated by depressive symptoms. However, there is no evidence directly examining the neural mechanisms of learning in individuals with TBI with and without depression. The proposed research explores this distinction.

The elucidation of the neural mechanisms associated with learning in individuals with TBI with and without clinical depression will inform 1) scientific knowledge about the effect of depression on the injured brain, 2) TBI interventions about the effectiveness of feedback and its timing, and 3) interventions for other clinical populations that require rehabilitation and have high occurrence of depression. These objectives lie at the heart of the mission of the National Institute of Neurological Disorders and Stroke as they will broaden "fundamental knowledge about the brain and nervous system" associated with learning in TBI and the knowledge gained from fulfilling the above objectives will "reduce the burden" of learning deficits after TBI.

To test these hypotheses, participants will be recruited based on structured clinical interview performed by the team member trained in psychiatric interviewing. Qualified participants will perform an experiment during which they will first study word pairs outside of the functional magnetic resonance imaging scanner. Then, in the scanner, participants will see word pairs again in a multiple-choice format and will have to choose a match for each word. After participants make their choice, feedback will be presented either immediately or after a delay of 25 minutes. The experiment will end with the Test phase, which takes place outside of the scanner, where participants will be presented with the words in the multiple-choice format again so the influence of each feedback type on learning can be evaluated.

Investigators hypothesize that depressed individuals with and without TBI will learn better from delayed compared to immediate feedback, because learning through delayed feedback relies on a different neural mechanism, which is not affected by depression and TBI, compared to learning through immediate feedback. Non-depressed individuals without TBI and clinically depressed individuals without TBI will also be recruited to delineate the influences of depression from the impact of TBI on the brain.

ELIGIBILITY:
Inclusion Criteria:

* I am between the ages of 18 and 65.
* I have been diagnosed with a TBI.
* I am an individual without TBI.
* I am right-handed.
* I have normal vision or corrected to normal vision.
* I can read and speak English fluently.
* I do or do not have a current diagnosis of Depression.
* I am not currently pregnant.

Exclusion Criteria:

* I have had a neurological disease, other than TBI.
* I have a significant history of alcohol or drug abuse as determined by study staff.
* I have metal in my body (shrapnel, piercing that cannot be taken off, retainer on the upper jaw).
* I have something in my body that restricts me from having an MRI such as: an aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or auto-defibrillator; cochlear implant (internal hearing aids); ocular foreign body (e.g. metal shavings in my eye), insulin pump or any pre- existing eye conditions (such as blurry vision, seeing double, and abnormal eye movements).
* I experience discomfort in closed spaces (claustrophobia).
* I have been diagnosed with a neurologic illness such as epilepsy, brain tumors, etc. (e.g. schizophrenia and bipolar disorder).
* I have had corticosteroid treatment less than a month ago as determined by study staff review of my medications.
* I have been informed by my doctor that is it unsafe for me to receive regular MRI as part of my medical care.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Learning accuracy | Collected during the single 1 day study
  Participants' learning accuracy (in percent) assessed with Eprime software
functional MRI | Collected during the single 1 day study
  Participants brain activity

SECONDARY OUTCOMES:
Verbal Paired Associates test | Collected during the single 1 day study
  Verbal learning and memory assessment
Logical Memory test | Collected during the single 1 day study
  Verbal learning and memory assessment
Delis-Kaplan Executive Function System | Collected during the single 1 day study
  Executive functioning assessment
Test of Premorbid Functioning | Collected during the single 1 day study
  Pre-morbid cognitive and memory functioning assessment
Ruff 2 & 7 Selective Attention Test | Collected during the single 1 day study
  Attention Assessment
Wechsler Adult Intelligence Scale, 4th edition | Collected during the single 1 day study
  Working memory/processing assessment
Behavioral Inhibition/Behavioral Approach Scale | Collected during the single 1 day study
  Questionnaire
GAD | Collected during the single 1 day study
  Questionnaire
PCL | Collected during the single 1 day study
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Dobryakova, PHD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No